CLINICAL TRIAL: NCT00548782
Title: Paleolithic Diets and Metabolic Control in Type 2 Diabetes Mellitus
Brief Title: Paleolithic Diets vs T2D and Improvements in the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H84763129001
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Paleolithic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Subjects will be placed on Paleolithic diet and markers of insulin resistance, lipid profiles and vascular reactivity will be measured. a paleolithic diet excludes dairy, grains, legumes and processed foods.
  Interventions: Other: Paleolithic diet
- B (Active Comparator): Subjects will be placed on ADA ( American Diabetes Association) recommended diet and markers of insulin resistance, lipid profiles and vascular reactivity will be measured. An ADA diet is lower fat and more whole grains.
  Interventions: Other: ADA ( American Diabetes Association) recommended diet

INTERVENTIONS:
Other: Paleolithic diet — diet
  Arms: A
Other: ADA ( American Diabetes Association) recommended diet — diet
  Arms: B

SUMMARY:
This study proposes to evaluate the physiological effects of eating Paleolithic type diet ("hunter-gatherer's diet") on Type 2 diabetic patients. The diet essentially consists of fruits, vegetables, nuts, lean meats, excludes dairy products and grains.Subjects will be randomized into taking either ADA (American Diabetic Association) recommended diet or Paleolithic diet for 21 days. The research kitchen will provide all food items and total calories in both groups will be adjusted to maintain baseline weight. Blood and urine test will be done in the first 3 days, last 3 days and 1 month after the study period to study and compare the effects of the two diets on subjects glucose control, lipid profile and other parameters of cardiovascular physiology.

We hypothesize that a palaeolithic diet in subjects with Type 2 diabetes mellitis, will result in improvement in above parameters and lead to improvement in glucose control with less need for diabetes medicines (either lower doses or fewer medications) to a greater extent than in subjects fed with ADA diet, without any change in weight. We also expect a beneficial effect on blood vessel function, lipid profiles and blood pressure.

DETAILED DESCRIPTION:
This study proposes to evaluate the physiological effects of eating Paleolithic type diet ("hunter-gatherer's diet") on Type 2 diabetic patients. The diet essentially consists of fruits, vegetables, nuts, lean meats, excludes dairy products and grains.Subjects will be randomized into taking either ADA (American Diabetic Association) recommended diet or Paleolithic diet for 21 days. The research kitchen will provide all food items and total calories in both groups will be adjusted to maintain baseline weight. Blood and urine test will be done in the first 3 days, last 3 days and 1 month after the study period to study and compare the effects of the two diets on subjects glucose control, lipid profile and other parameters of cardiovascular physiology.

We hypothesize that a palaeolithic diet in subjects with Type 2 diabetes mellitis, will result in improvement in above parameters and lead to improvement in glucose control with less need for diabetes medicines (either lower doses or fewer medications) to a greater extent than in subjects fed with ADA diet, without any change in weight. We also expect a beneficial effect on blood vessel function, lipid profiles and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Age >= 18 yrs
* BMI < 40 kg/m2
* Normal cardiac, renal and hepatic function

Exclusion Criteria:

* Subjects on thiazolidinediones ( Avandia, Actos) or other medications that interfere with the testing procedures
* Subjects unwilling or unable to follow the diet specified
* Pregnant women
* Subjects who are unable to understand the consent form
* Hematocrit less than 30
* Patients with defibrillators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2013-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
decreased insulin secretion | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Franca Angeli, MD, Principal Investigator — University of California, San Francisco; Umesh Masharani, MRCP, Principal Investigator — University of California, San Francisco; Lynda Frassetto, MD, Principal Investigator — University of California, San Francisco; Shelley MCCoy, Study Director — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No